CLINICAL TRIAL: NCT00374231
Title: A Single Center, Pilot Study of Corticosteroid Discontinuation in Liver Transplant Recipients Utilizing a Tacrolimus/Mycophenolate Mofetil Based Maintenance Immunosuppression Protocol
Brief Title: Single Center Pilot Study of Corticosteroid Discontinuation in Liver Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, E. Steve Woodle, MD, FACS, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSWD Liver
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Results first posted 2015-12-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-11

CONDITIONS: Liver Transplantation
Keywords: Liver; Transplant; Corticosteroid withdrawal; Tacrolimus; CellCept; MMF; Mycophenolate mofetil
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Immunosuppression (Experimental): All the patients who enroll in this study will receive the same medications (tacrolimus, mycophenolate mofetil, and a short course of steroids) to prevent rejection of the liver transplant. All participants will be gradually taken off prednisone if they are 90 days or longer post liver transplant and have not had a rejection in the last 30 days.
  Interventions: Drug: tacrolimus; Drug: mycophenolate mofetil; Drug: Prednisone

INTERVENTIONS:
Drug: tacrolimus — Tacrolimus is a pill taken orally. Dose, frequency and duration will be decided by the study doctor on a case-by-case basis.
  Other Names: Prograf, FK506
Drug: mycophenolate mofetil — Mycophenolate mofetil is a pill taken orally. Dose, frequency and duration will be decided by the study doctor on a case-by-case basis.
  Other Names: MMF, CellCept
Drug: Prednisone — Prednisone is a pill taken orally. Dose, frequency and duration will be decided by the study doctor on a case-by-case basis.
  Other Names: corticosteriods

SUMMARY:
To determine the safety and efficacy of early corticosteroid discontinuation in liver transplant recipients more than 90 days post transplant, utilizing a combination of two drugs (tacrolimus and mycophenolate mofetil) for maintenance immunosuppressant therapy.

DETAILED DESCRIPTION:
To determine the safety and efficacy of early corticosteroid discontinuation in liver transplant recipients more than 90 days post transplant, utilizing a combination of two drugs (tacrolimus and mycophenolate mofetil) for maintenance immunosuppression therapy.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 90 days post transplant.
* Free from rejection within the last 30 days.
* Patient with primary diagnosis of AIH will be evaluated on an individual basis.
* Negative pregnancy test.
* Practicing an acceptable method of birth control.
* Capable of providing written informed consent.

Exclusion Criteria:

* Rejection within the last 30 days.
* Patients with AIH unable to discontinue corticosteroids.
* Patients currently receiving systemic corticosteroids for other medical diseases in which the physician feels discontinuation is contraindicated.
* Known sensitivity or contraindication to tacrolimus or MMF.
* Kidney, pancreas, islet, heart, lung, or small bowel transplant recipient.
* Pregnant or lactating.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Woodle, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 3/2003 to 11/2005 forty adult deceased donor liver transplant recipients were enrolled. Subjects were eligible once they were greater than 90 days post liver transplant provided they had a 30 day rejection free period prior to enrollment.
Groups:
- Corticosteroid Withdrawal: Discontinue prednisone at 90 days or longer post liver transplant if rejection free previous 30 days.
Period: Overall Study
Arm/Group | Corticosteroid Withdrawal
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Tacrolimus and Mycophenolate Mofetil: All the patients who enroll in this study will receive the same medications (tacrolimus, mycophenolate mofetil, and a short coarse of steroids) to prevent rejection of the liver transplant. All participants will be gradually taken off prednisone if they are 90 days or longer post liver transplant and have not had a rejection in the last 30 days.
  tacrolimus : Tacrolimus is a pill taken orally. Dose, frequency and duration will be decided by the study doctor on a case-by-case basis.
  mycophenolate mofetil : Mycophenolate mofetil is a pill taken orally. Dose, frequency and duration will be decided by the study doctor on a case-by-case basis.
Arm/Group | Tacrolimus and Mycophenolate Mofetil
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 36
  More than one race | 0
  Unknown or Not Reported | 0
Cause of Liver Disease [Number; unit: participants]
  Alcoholic Liver Disease | 9
  Viral Hepatitis C | 6
  Primary Schlerosing Cholangitis | 6
  Hepatocellular Carcinoma | 6
  Cryptogenic Cirrhosis | 6
  Non-alcholic Steatohepatitis | 2
  Autoimmune Hepatitis | 1
  Other | 4

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Biopsy Confirmed Acute Rejection at 12 Months.
Time Frame: 12 months
Measure: Number; unit: participants
Groups:
- Corticosteroid Withdrawa.: All the patients who enroll in this study will receive the same medications (tacrolimus, mycophenolate mofetil, and a short coarse of steroids) to prevent rejection of the liver transplant. All participants will be gradually taken off prednisone if they are 90 days or longer post liver transplant and have not had a rejection in the last 30 days.
  tacrolimus: Tacrolimus is a pill taken orally. Dose, frequency and duration will be decided by the study doctor on a case-by-case basis.
  mycophenolate mofetil: Mycophenolate mofetil is a pill taken orally. Dose, frequency and duration will be decided by the study doctor on a case-by-case basis.
Arm/Group | Corticosteroid Withdrawa.
Number analyzed (Participants) | 40
participants | 5

2. Secondary Outcome: Patient Survival.
Time Frame: 12 months
Measure: Number; unit: participants
Groups:
- Corticosteroid Withdrawal: All the patients who enroll in this study will receive the same medications (tacrolimus, mycophenolate mofetil, and a short coarse of steroids) to prevent rejection of the liver transplant. All participants will be gradually taken off prednisone if they are 90 days or longer post liver transplant and have not had a rejection in the last 30 days.
  tacrolimus: Tacrolimus is a pill taken orally. Dose, frequency and duration will be decided by the study doctor on a case-by-case basis.
  mycophenolate mofetil: Mycophenolate mofetil is a pill taken orally. Dose, frequency and duration will be decided by the study doctor on a case-by-case basis.
Arm/Group | Corticosteroid Withdrawal
Number analyzed (Participants) | 40
participants | 39

3. Other Pre Specified Outcome: Time Post Transplant Corticosteroid Withdrawal
Description: The mean days from post transplant corticosteroid withdrawal.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Corticosteroid Withdrawal
Number analyzed (Participants) | 40
days | 257 (511)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Tacrolimus and Mycophenolate Mofetil
Serious Adverse Events (participants affected / at risk) | 9/40
Other Adverse Events (participants affected / at risk) | 3/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus and Mycophenolate Mofetil (N=40)
Lower Extremity Cellulites (Infections and infestations) | 1 (1)
Acute Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Portal Vein Stenosis (Vascular disorders) | 2 (2)
Total Knee Anthroplasty (Vascular disorders) | 1 (1)
Incisional Hernia Repair (Skin and subcutaneous tissue disorders) | 1 (1)
Lymphocele (General disorders) | 1 (1)
Moderate Allograft Rejection (Renal and urinary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus and Mycophenolate Mofetil (N=40)
Allograft rejection (mild) (Renal and urinary disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes